CLINICAL TRIAL: NCT02692794
Title: Large Scale Cerebral Oximetry During Sinus Endoscopy
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: GCO 15-1192
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Endoscopic Sinus Surgery; Chronic Rhinosinusitis
Keywords: sinusitis; oximetry; paranasal sinus diseases
MeSH Terms: conditions — Sinusitis; Paranasal Sinus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Specify all types of biospecimens to be retained (e.g., whole blood, serum, white cells, urine, tissue)
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Deliberate hypotension, reverse Trendelenburg position, and hyperventilation are techniques utilized during functional endoscopic sinus surgery to attempt to reduce surgical bleeding. These methods reduce blood flow to the head and neck area and assist in reducing bleeding during surgery but they may predispose patients to cerebral ischemia. Large scale studies necessary to conduct adequate statistical analysis regarding the effect of cerebral oximetry on otolaryngology surgery has not been extensively studied. This study seek to address the question of whether cerebral oximetry in the FESS population can help evaluate major and minor post operative morbidity, as well as the quality of recovery from surgery. Cerebral oximeters are small, noninvasive stickers applied to the forehead of participants and give the examiners data regarding the level of oxygen saturation around the brain during the course of surgery. During the course of such procedures, where blood flow to the head and neck area is intentionally decreased to assist in reducing bleeding during surgery, the levels of oxygen saturation around the brain may pose as a predictor or major and minor post operative morbidity, as well as the quality of recovery from surgery. Outcome measures will include major post operative complications, such as neurological and cardiac complications, and minor post operative morbidity, such as length of post anesthesia care unit (PACU) length of stay, nausea, and vomiting. Quality of recovery will also be assessed using a survey conducted in the PACU and again at the first post operative visit approximately one week after surgery.

DETAILED DESCRIPTION:
Research Plan

This study will be conducted at Mount Sinai Hospital. Patients will be recruited by reading the operating room schedule in advance and contacting patients over the phone to explain the study, risks and benefits, and obtain informed consent prior to admission to the hospital.

Objective 1 The specific aim of this observational study is to evaluate changes in cerebral tissue oxygen saturation in patients undergoing head and neck surgery under general anesthesia with mechanical ventilation using the Casmed Foresight cerebral oximeter.

Ensuring patient safety in surgeries upon the head and neck is a complex task in anesthesiology. These patients present a myriad of concerns that need to be considered to create a safe and thorough anesthetic plan that include potentially difficult airways, varied patient positioning, and the intricate involvement of anesthetic drugs upon the quality of the surgical field. During common procedures such as sinus endoscopy, patients undergo endotracheal intubation and mechanical ventilation for airway protection and a strategy of deliberate hypotension is implemented with the goal of creating a clean surgical field that minimizes avoidable bleeding. The objective of this strategy is to allow the surgeons to complete their procedure more quickly and with less hypothetical risk of injury due to poor visualization of structures. However, this strategy of deliberate hypotension carries with it the potential risk of cerebral hypoperfusion as the lower limits of cerebral autoregulation are not known on an individual patient basis. Furthermore, mechanical ventilation- particularly with hyperventilation- can further decrease cerebral blood flow and potentially compromise cerebral perfusion. The current standard of care to monitor the hemodynamics of patients undergoing these procedures are standard American Society of Anesthesiologists monitors, which includes non-invasive blood pressure measurements. The investigators propose the use of a non-invasive monitor of cerebral oxygenation with cerebral oximeter probes in a prospective, observational study of a series of patients undergoing routine head and neck surgery.

ELIGIBILITY:
Inclusion Criteria:

- patients undergoing elective head and neck surgery at Mount Sinai Hospital in which 1) the patient will be intubated and mechanically ventilated, with 2) head of bed elevated, and in which 3) an anesthesiologist could consider deliberate hypotension as part of their management

Exclusion Criteria:

* patients under 18 years old
* patients who are currently prisoners
* patients who do not appear to have capacity to consent to the study
* patients who cannot provide informed consent in English
* pregnant women
* patients who decline to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing primary or revision endoscopic sinus surgery for chronic rhinosinusitis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-10; Primary Completion 2016-06-20 (Actual); Study Completion 2016-06-20 (Actual)

PRIMARY OUTCOMES:
Post-operative Quality of Recovery Scale | Day 1- 1 hour post-operatively
  Post-operative Quality of Recovery Scale to assess cognitive delay in patients undergoing sinus surgery
Post-operative Quality of Recovery Scale | Day 2
  Post-operative Quality of Recovery Scale to assess cognitive delay in patients undergoing sinus surgery

SECONDARY OUTCOMES:
Incidence of nausea/vomiting | Day 1 - 1 hour post-operatively
  Increased incidence of nausea/vomiting post-operatively in patients with cerebral desaturation during the course of sinus surgery

OTHER OUTCOMES:
Incidence of pain experience | Day 1 - 1 hour post-operatively
  Incidence of post-operative pain experienced in patients with cerebral desaturation during the course of sinus surgery

CONTACTS AND LOCATIONS:
Overall Officials: Satish Govindaraj, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No